CLINICAL TRIAL: NCT05434650
Title: Abbott Atrial Fibrillation Post Approval Study
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10436
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Arrhythmia; Atrium; Fibrillation; Atrial Tachycardia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treatment group: Single arm group to receive ablation
  Interventions: Device: electrophysiology study and ablation with an Abbott Ablation Catheter

INTERVENTIONS:
Device: electrophysiology study and ablation with an Abbott Ablation Catheter — During the cardiac ablation procedure, an ablation catheter (a thin, flexible tube that can be threaded through the blood vessels to the heart) will deliver radiofrequency energy (a type of heat) to one or more areas in the upper left chamber of the heart that is causing the irregular heartbeat. The tip of the catheter will transmit energy to one or more small spots of heart tissue. This energy creates a small scar on the heart. This scar will block the electrical pathway that is causing the rapid heartbeat

SUMMARY:
This post-approval study is designed to provide continued real-world clinical evidence to confirm the safety and long-term effectiveness of atrial fibrillation (AF) radiofrequency (RF) technologies (e.g. TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE)) for the treatment of AF.

DETAILED DESCRIPTION:
This post-approval study is a prospective, non-randomized, single arm, multicenter, observational study to evaluate the continued safety and effectiveness of AF RF technologies, including the TactiCath SE. The primary effectiveness endpoint will be the proportion of subjects with freedom from AF recurrence after the initial catheter ablation procedure through 12 months of follow-up (includes a 90-day blanking period). Secondary effectiveness endpoints will be the proportion of subjects with freedom from AF recurrence after the initial catheter ablation procedure through 24 and 36 months of follow-up (includes a 90-day blanking period). The acute primary safety endpoint will be the rate of device and/or procedure-related serious adverse events (SAE) with onset within 7-days of the index ablation procedure utilizing the study catheter. The secondary, long-term safety endpoint will be the rate of device and/or procedure-related SAEs from the index ablation procedure. An independent Clinical Event Committee (CEC) will review all Adverse Device Effects (ADEs) and SAEs and will adjudicate causality relative to the primary safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation-related procedure.
2. Documented symptomatic persistent AF, which is defined as continuous AF sustained beyond 7 days and less than 1 year that is documented by a physician's note AND one of the following:

   1. a 24-hour Holter within 180 days prior to consent/enrollment, showing continuous AF OR
   2. two electrocardiograms (from any form of rhythm monitoring) showing continuous AF:

   i. that are taken at least 7 days apart but less than 12 months apart. ii. If electrocardiograms are more than 12 months apart, there must be one or more SR recordings in between or within 12 months prior to consent/enrollment NOTE: The most recent ECG must be within 180 days of consent/enrollment. Documented evidence of the AF episode must either be continuous AF on a 12-lead ECG or include at least 30 seconds of AF from another ECG device.
3. Subject must have failed, intolerance, or contraindication to a Class I-IV AAD medication.
4. Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

1. Previously diagnosed continuous AF >12 months (longstanding persistent AF)
2. Previous left atrial surgical or catheter ablation for atrial fibrillation or a previous procedure that required an incision in the left atrium with resulting scar
3. Documented or known intracardiac thrombus on imaging
4. History of atriotomy or ventriculotomy within 4 weeks prior to the initial procedure
5. Patients with prosthetic valves
6. Diagnosed atrial myxoma
7. Acute illness or active systemic infection or sepsis
8. Patient is unlikely to survive the protocol follow up period of 36 months
9. Presence of other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
10. Enrollment in an investigational study evaluating another device, biologic, or drug that may interfere with this clinical investigation at the time of the initial procedure or within 30 days prior to the initial procedure
11. Investigator deems at the time of screening for inclusion in the study that the patient's treatment plan does not or likely will not include use of the study catheter

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This clinical investigation will enroll subjects of all genders who have drug refractory, symptomatic, persistent AF.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with freedom from AF recurrence post 90-day blanking period at 12 months | 12 months
  AF recurrence is defined as:
  1. Documented AF/atrial flutter (AFL)/atrial tachycardia (AT) episodes of > 30 seconds duration following the blanking period
  2. Repeat ablation for AF/AFL/AT following the blanking period
  3. Cardioversion (electrical or pharmaceutical) for the treatment of AF following the blanking period
  4. A new Class I/III AAD or a previously failed Class I/III AAD at a dose greater than the highest historical dose for AF is needed following the blanking period
Rate of device and/or procedure-related serious adverse events (SAE) with onset within 7-days of the index ablation procedure | 7 days
  Device and/or index procedure-related SAEs are defined below:
  * Atrio-esophageal fistula
  * Cardiac tamponade/perforation
  * Death
  * Heart block
  * Myocardial infarction (MI)
  * Pericarditis
  * Phrenic nerve injury resulting in diaphragmatic paralysis
  * Vagal nerve injury/gastroparesis
  * Pulmonary edema (respiratory insufficiency)
  * Pulmonary vein stenosis
  * Stroke/cerebrovascular accident (CVA)
  * Thromboembolism
  * Transient ischemic attack
  * Vascular access complications (including major bleeding events3)

SECONDARY OUTCOMES:
the proportion of subjects with freedom from AF recurrence post 90-day blanking period at 24 months and 36 months | 36 months
  AF recurrence is defined as:
  1. Documented AF/atrial flutter (AFL)/atrial tachycardia (AT) episodes of > 30 seconds duration following the blanking period
  2. Repeat ablation for AF/AFL/AT following the blanking period
  3. Cardioversion (electrical or pharmaceutical) for the treatment of AF following the blanking period
  4. A new Class I/III AAD or a previously failed Class I/III AAD at a dose greater than the highest historical dose for AF is needed following the blanking period
the rate of device and/or procedure-related SAEs from the index ablation procedure, descriptively evaluated at 12 months, 24 months, and 36 months | 36 months
  Device and/or index procedure-related SAEs are defined below:
  * Atrioesophageal fistula
  * Cardiac tamponade/perforation
  * Death
  * Heart block
  * Myocardial infarction (MI)
  * Pericarditis
  * Phrenic nerve injury resulting in diaphragmatic paralysis
  * Pneumothorax
  * Pulmonary edema (respiratory insufficiency)
  * Pulmonary vein stenosis
  * Stroke/cerebrovascular accident (CVA)
  * Thromboembolism
  * Transient ischemic attack
  * Vascular access complications (including major bleeding events)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, Study Director — Abbott
Locations (20):
- United States (20):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Arkansas Cardiology, Little Rock, Arkansas
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sequoia Hospital, Redwood City, California
  - Northside Hospital, Atlanta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Providence Hospital, Southfield, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Patrick Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oklahoma Heart Hospital South, Oklahoma City, Oklahoma
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Methodist Hospital of San Antonio, San Antonio, Texas
  - St. Marks Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Chippenham Hospital, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided